CLINICAL TRIAL: NCT05927298
Title: Province of Ontario Strategy for Personalized Management of Pancreatic Cancer Trial
Acronym: ProsperPanc
Status: Recruiting | Type: Observational
Sponsor: University Health Network, Toronto (Other)
Collaborators: Ontario Institute for Cancer Research (Other); Ottawa Hospital Research Institute (Other); London Health Sciences Centre Research Institute OR Lawson Research Institute of St. Joseph's (Other)
Responsible Party: Sponsor
Other Study IDs: OZUHN-011
Record Dates: First submitted 2023-01-25; First posted 2023-07-03 (Actual); Last update posted 2024-10-15 (Actual); Status verified 2024-10

CONDITIONS: Pancreas Cancer
MeSH Terms: conditions — Pancreatic Neoplasms

STUDY DESIGN:
Observational Model: Cohort | Time Perspective: Prospective
Biospecimen Retention: Samples With DNA — Tumour tissue will undergo WGS/RNAseq. Germline blood samples will be used as reference
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

GROUPS / COHORTS (2):
- Cohort 1: Upfront resectable PDAC
  Interventions: Other: Non-interventional
- Cohort 2: Advanced (unresectable PDAC or metastatic)
  Interventions: Other: Non-interventional

INTERVENTIONS:
Other: Non-interventional — Standard of care intervention

SUMMARY:
This is a prospective, multi-centre, translational and observational study. Two cohorts of patients with pancreatic ductal adenocarcinoma (PDAC) are eligible to enroll 1) Upfront resectable PDAC 2) Advanced (unresectable PDAC or metastatic). Patients will have tissue either at resection or from a biopsy at enrolment processed for whole genome sequencing, RNA sequencing and for establishment of patient derived organoids (PDOs). Background epidemiological history and outcome data will be prospectively annotated. Serial blood and stool samples will be collected for exploratory analyses. All electronic medical record information will also be collected. Data will be used to determine if an integrated correlative analysis of whole genome sequencing/RNAsequencing (WGS/RNAseq) and PDOs in the enrolled population will increase the number of patients receiving a precision-matched treatment in Ontario

DETAILED DESCRIPTION:
This study is being done to answer the following question: Can creating 3D models using tumour samples and looking at genetic information from pancreatic ductal adenocarcinoma (PDAC) tumours, help us to provide more patients with a specific, personalized treatment? Two groups of patients with PDAC are eligible to enroll 1) PDAC patients that will go straight to surgery 2) PDAC patients where the disease is either too advanced for a surgical option, or the disease has spread to other areas in the body. Patients will have tumour tissue taken either during their surgery or from a biopsy at enrolment. Background history, outcome data, questionnaires, series of blood draws and stool samples will be collected for analyses. All electronic medical record information will also be collected.

Researchers are looking for better ways of understanding and treating pancreatic cancer by looking to see how useful it is to know about changes and characteristics in the genes in the tumour (molecules that contain instructions for the development and functioning of the cells). Results from analyzed data may be useful in choosing treatments for enrolled patients and for patients in the future. Patients current treatment plan will not change if they choose to take part in this study.

ELIGIBILITY:
Inclusion Criteria:

1. Patients must have either upfront resectable PDAC or advanced (unresectable or metastatic) PDAC (borderline PDAC and those planned for neoadjuvant chemotherapy excluded)
2. Patients with a histological or radiological diagnosis of pancreatic ductal adenocarcinoma (PDAC). For patients awaiting histological confirmation, tissue obtained at study enrolment or can suffice. For those patients who undergo a resection, surgical tissue will be used.
3. For patients enrolling with resectable PDAC (cohort 1) - the definition of resectability will be according to NCCN guidelines and the patient must be planned for a surgery first approach.
4. For patients with advanced PDAC (cohort 2), all stages are eligible including locally advanced unresectable, first-line metastatic, second-line (or beyond) metastatic.
5. In advanced PDAC patients (cohort 2) where a single lesion is to be biopsied, the lesion should be amenable to a core needle biopsy as judged by a staff radiologist. A minimum of 4 to 6 x 18 Gauge (G) good quality tumour cores must be safely obtainable under CT or US guidance.
6. Patients must have a life expectancy of ≥ 6 months
7. ECOG 0-1
8. Patient must be suitable for systemic therapy
9. Patients should have organ function deemed sufficiently adequate to receive systemic therapy

Exclusion Criteria:

1. Certain histologies are excluded: colloid, high grade neuroendocrine;
2. For patients enrolling in cohort 2 - Patients without a tumour lesion amenable to biopsy or with tumour lesions that are not safe for sampling a minimum of 4 to 6 x 18G good quality tumour cores by image guided core needle biopsy as judged by a staff radiologist.
3. Patients who are not fit enough to undergo a tumour biopsy for any reason as judged by the investigator; this includes patients who cannot stop anticoagulation therapy.
4. For cohort 1 - patients receiving neoadjuvant chemotherapy are excluded, (neoadjuvant immunotherapy is permitted)

Min Age: 18 Years | Sex: All
Age Groups: Adult, Older Adult
Study Population: 1. Upfront resectable PDAC not receiving neoadjuvant chemotherapy (Immunotherapy only regimens are eligible)
  2. Advanced (unresectable or metastatic) PDAC suitable for systemic therapy.
Sampling Method: Non-Probability Sample
Enrollment: 200 (Estimated)
Dates: Start 2023-03-06 (Actual); Primary Completion 2027-03-06 (Estimated); Study Completion 2027-03-06 (Estimated)

PRIMARY OUTCOMES:
Precision-Matched Treatment Utilization Rate | 4 years
  Number of patients receiving precision-matched treatment in Ontario based on integrated correlative analysis of whole-genome sequencing (WGS), RNA sequencing (RNAseq), and patient-derived organoids (PDOs).

SECONDARY OUTCOMES:
Build a comprehensive dataset of pancreatic cancer specimens (tissue and blood) and matched patient-derived organoids (PDOs) | 4 years
Correlate drug sensitivities in patient-derived organoids (PDOs) and molecular information | 4 Years
Correlate immune phenotypes and molecular profiles | 4 Years

OTHER OUTCOMES:
Develop an electronic medical record (EMR) platform utilizing artificial intelligence (AI) modeling | 4 Years
Correlate serial plasma whole-genome sequencing (WGS) and tissue WGS | 4 Years
Characterize the epigenome in established patient-derived organoids (PDOs) | 4 Years
Assess oncolytic virus efficacy in combination with immune checkpoint inhibitors in a subset of 50 patient-derived organoids (PDOs) co-cultured with autologous peripheral blood mononuclear cells (PBMCs) | 4 Years
Identify microbiome differences in patients at various stages of pancreatic ductal adenocarcinoma (PDAC) and their correlation with whole-genome sequencing (WGS)/RNA subtypes | 4 Years
Document stroma subtypes in pancreatic cancer and their correlation with clinical outcomes | 4 Years
Evaluate treatment responses in patients receiving precision-matched treatment using the Response Evaluation Criteria in Solid Tumors (RECIST) version 1.1 | 4 Years
Investigate the involvement of genetic and environmental factors in the development and progression of pancreatic cancer | 4 Years
Assess comparability between WGS and commercial panel | 4 Years
Explore the feasibility and efficacy of utilizing digitized whole-slide images of biopsy or resection specimens for an AI-based digital pathology prediction system | 4 Years

CONTACTS AND LOCATIONS:
Overall Officials: Erica Tsang, MD, Principal Investigator — University Health Network, Toronto
Locations (1):
- Princess Margaret Cancer Centre, Toronto, Ontario, Canada

IPD SHARING:
Plan to Share IPD: No